CLINICAL TRIAL: NCT07167082
Title: Hospitalized Cancer Patients: Prognostic Value of Hand Grip Strength - A Prospective Cohort Study
Brief Title: Hand Grip Strength and Prognosis in Hospitalized Cancer Patients
Acronym: PRO-HAND
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Department of Medical Oncology, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-1105; AEŞH-BADEK-2024-1105 (Other: Ankara Etlik City Hospital Ethics Committee)
Record Dates: First submitted 2025-08-23; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Hospitalizations; Sarcopenia; Cachexia; Cancer; Sarcopenia
Keywords: Hand Grip Strength; Prognosis; Hospitalized Cancer Patients; Cachexia; Malnutrition; Functional Decline; Mortality
MeSH Terms: conditions — Neoplasms; Sarcopenia; Cachexia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized Cancer Patients: This cohort consists of adult patients (aged 18-80 years) with pathologically confirmed cancer who are admitted to the hospital for at least 48 hours. Hand grip strength is measured within the first 24 hours of admission using a standardized dynamometer protocol. Patients are followed prospectively for 30 days to evaluate primary and secondary outcomes including all-cause mortality, functional decline, hospital stay duration, readmission, and major complications.
  Interventions: Other: Hand Grip Strength Measurement

INTERVENTIONS:
Other: Hand Grip Strength Measurement — Hand grip strength will be measured within the first 24 hours of hospitalization using a calibrated hand dynamometer. Measurements will be performed on the dominant hand, with patients seated, following standardized international procedures. Three consecutive measurements will be obtained, and the average value will be recorded. The test is non-invasive, quick, and performed by oncology clinicians trained in the protocol.

SUMMARY:
This prospective cohort study aims to investigate the relationship between hand grip strength and prognosis in hospitalized cancer patients. Hand grip strength, a simple, rapid, and non-invasive measure of overall muscle function, is increasingly recognized as an indicator of frailty, nutritional status, and physical health. The study will evaluate whether lower hand grip strength is associated with higher short-term mortality (30-day all-cause mortality) and adverse clinical outcomes, including ICU admission, hospital readmission, and functional decline.

DETAILED DESCRIPTION:
Hand grip strength declines with age and is associated with frailty, sarcopenia, and cancer cachexia. It is a reliable prognostic marker in cancer patients. In this prospective cohort study, hospitalized patients with pathologically confirmed cancer will undergo hand grip strength measurement within the first 24 hours of admission using a calibrated hand dynamometer. Measurements will be performed on the dominant hand, with patients seated, following international standardized procedures. Three consecutive measurements will be obtained, and the average value will be recorded. Assessments will be conducted by oncology clinicians trained in the protocol. Patients will be followed for 30 days to evaluate primary and secondary endpoints, including all-cause mortality, functional decline, length of hospital stay, intensive care unit admission, readmission, and major complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Pathologically confirmed diagnosis of cancer
* Hospitalized with an expected hospital stay of more than 48 hours
* Ability to provide written informed consent

Exclusion Criteria:

* Diagnosis of anorexia nervosa
* Acute pancreatitis or acute liver failure at admission
* History of gastric bypass surgery
* Presence of chronic active infections
* History of solid organ transplantation
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older with pathologically confirmed cancer who are admitted to the Ankara Etlik City Hospital, Department of Medical Oncology. Eligible participants are hospitalized for more than 48 hours and undergo hand grip strength measurement within 24 hours of admission. Patients represent a heterogeneous group of solid tumor cases across different cancer types and stages, reflecting a real-world hospitalized oncology population.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
30-day All-Cause Mortality | 30 days after hospital admission
  All-cause mortality within 30 days of hospital admission among cancer patients (Yes/No). Mortality status will be assessed through hospital records and follow-up. Hand grip strength values will be analyzed in relation to mortality risk.

SECONDARY OUTCOMES:
Intensive Care Unit Admission | 30 days after hospital admission
  Number of patients requiring ICU admission within 30 days of hospital admission (Yes/No).
Hospital Readmission | 30 days after discharge
  All-cause hospital readmission within 30 days of discharge (Yes/No).
Functional Decline - ECOG Performance Status | Baseline and 30 days after hospital admission
  Decline in functional status assessed by the Eastern Cooperative Oncology Group (ECOG) Performance Status (range 0-4; 0 = fully active, 1 = restricted in strenuous activity, 2 = ambulatory but unable to work, 3 = limited self-care, 4 = completely disabled; higher score = worse performance), comparing baseline and 30-day follow-up.
Length of Hospital Stay | Through initial hospitalization, up to 30 days
  Duration of initial hospitalization, measured in days from admission to discharge.
Major Complications | 30 days after hospital admission
  Incidence of major complications including hospital-acquired infection, respiratory failure, cardiovascular events, acute renal failure, or gastrointestinal failure within 30 days (Yes/No).
Functional Decline - Patient-Generated Subjective Global Assessment (PG-SGA) | Baseline and 30 days after hospital admission
  Decline in nutritional status assessed by the Patient-Generated Subjective Global Assessment (PG-SGA) Score (range 0-35; 0-1 = no intervention required, 2-3 = patient/family education, 4-8 = requires dietitian intervention, ≥9 = critical need for nutritional intervention and/or symptom management; higher score = worse nutritional status), comparing baseline and 30-day follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Medical Oncology Department, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No